CLINICAL TRIAL: NCT05395858
Title: REAL: A Pre-/Post-Intervention Descriptive Analysis and Cross-Sectional Survey to Evaluate Real-World Treatment Outcomes, Consumption, and Satisfaction With Damoctocog Alfa Pegol in US Hemophilia Treatment Centers
Brief Title: A Study to Learn More About Treatment With Damoctocog Alfa Pegol, How it is Used in Every Day Practice ("Real-World"), and How Satisfied People Who Receive Damoctocog Alfa Pegol Are in United States (US) Hemophilia Treatment Centers
Acronym: REAL
Status: Terminated | Type: Observational
Why Stopped: Bayer business decision to close the REAL study based on the following: Target objective of enrolling at least 20 patients into the retrospective part failed; Not enough available data that would be a meaningful addition to the literature.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21280
Record Dates: First submitted 2022-04-28; First posted 2022-05-27 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hemophilia A
Keywords: Bleeding disorder; Coagulation factor VIII; Blood Coagulation Disorders
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A patients: Patients will be identified via standard medical charts or electronic medical records (EMRs).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective analysis using database without any intervention assigned in the study.

SUMMARY:
People with hemophilia A do not have enough of a protein found naturally in the blood called "clotting factor 8", also known as FVIII. This protein helps the blood to clump together to prevent and stop bleeding. People with lower levels of FVIII or FVIII that does not work properly may bleed for a long time from minor wounds, bleed into their joints, or have internal bleeding.

The study treatment, Jivi (also called damoctocog alfa pegol), is already available as a treatment for people aged 12 years and older with hemophilia A, to help prevent bleeding, also known as "prophylactic" treatment. It works by replacing the missing FVIII, or the FVIII that does not work properly. It can also be used to stop bleeding that has already occurred and prior to surgery to prevent bleeding.

The main goal of this study is to learn how damoctocog alfa pegol is used in the "real world" as a treatment in the United States (US) and how well it works and what other treatments patients use while receiving damoctocog alfa pegol treatment. It will also determine how satisfied people are with the treatment. There will be no required visits with a study doctor in this study.

The study will include about 20 male or female patients in the US aged 12 years and over who have hemophilia A. All the patients in this study will have switched from their previous FVIII replacement treatment to damoctocog alfa pegol. While the patients are receiving damoctocog alfa pegol, they will complete a survey to say how they feel about the treatment. Their doctors will also record information about their treatment with damoctocog alfa pegol and how well it is working.

This study will collect information from the patients' medical records and surveys. They will use this information to find out more about treatment with damoctocog alfa pegol under "real world" conditions. They will look at:

* how often the patients receive damoctocog alfa pegol and how much they use
* what other treatments the patients received before receiving damoctocog alfa pegol, how they used it and how much they used
* how well damoctocog alfa pegol works at preventing bleeding, and how it compares to previous products used.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a diagnosis of hemophilia A
* Previously or currently treated with damoctocog alfa pegol for at least 6 months.
* Treated with damoctocog alfa pegol per the US approved label to include:

  * Aged ≥12 years at the time of damoctocog alfa pegol treatment initiation
  * Previously treated for hemophilia A with an FVIII replacement therapy other than damoctocog alfa pegol
  * Treatment modality of on-demand, prophylactic, intermittent prophylaxis or a combination thereof
* Have data in the medical record at the participating site as follows:

  * For a minimum of 6 months prior to the damoctocog alfa pegol initiation date
  * For a minimum of 6 months post-damoctocog alfa pegol initiation date AND the patient was receiving treatment with damoctocog alfa pegol during this 6-month follow-up period AND this data is dated prior to the central institutional review board (IRB) approval date for the study
  * To include the FVIII replacement therapy most recently received prior to the initiation of damoctocog alfa pegol
* For patients in the prospective cohort

  * Signed informed consent
  * Current treatment with damoctocog alfa pegol or discontinued use of damoctocog alfa pegol within 3 months prior to the date of enrollment into the retrospective cohort.

Exclusion Criteria:

* Diagnosis of any other bleeding/coagulation disorder other than hemophilia A.
* Participation in any past or current damoctocog alfa pegol interventional trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: United States patients aged ≥12 years diagnosed with hemophilia A (congenital FVIII deficiency) who switched from a previous FVIII replacement treatment to damoctocog alfa pegol. No investigational products will be administered in this study.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Frequency of damoctocog alfa pegol infusions | From index date through the date of central IRB approval (3 years and 8 months)
  Reported as infusions. IRB: institutional review board

SECONDARY OUTCOMES:
Descriptive summary of pre-damoctocog alfa pegol treatment regimen | 6 months prior to the index date.
Descriptive summary of damoctocog alfa pegol treatment regimen. | Up to 5 years from index date
Descriptive summary of post-damoctocog alfa pegol treatment regimen, if applicable. | Up to 4 years
  Only applicable for patients who discontinue damoctocog alfa pegol treatment regime.
Descriptive summary of changes in pre-damoctocog alfa pegol treatment regimes | 6 months prior to the index date.
Descriptive summary for reasons for treatment discontinuation of pre-damoctocog alfa pegol treatment regimes. | 6 months prior to the index date.
Annualized number of spontaneous, joint, and trauma bleeds before initiation of treatment with damoctocog alfa pegol. | 6 months prior to the index date.
Annualized number of spontaneous, joint, and trauma bleeds post initiation of treatment with damoctocog alfa pegol. | Up to 5 years from index date

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - Tulane University, New Orleans, Louisiana
  - Regents of the University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.